CLINICAL TRIAL: NCT03009331
Title: Descriptive and Comparative Study of Respiratory Function in the Postoperative Cardiac Surgery Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Martinsson, Medical Doctor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMartinssonthorax
Record Dates: First submitted 2016-12-14; First posted 2017-01-04 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Atelectasis
Keywords: Postoperative pulmonary dysfunction; Postoperative pulmonary complication; Recruitment manouver; Prone position
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Prone Position; Ventilators, Mechanical; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone position (Experimental): Intervention: Lungrecruitment in prone position. Device: Ventilator Flow-i, Peak inspiratory pressure 40 cmH2O, PEEP 20 cm H2O during 30 s.
  Interventions: Procedure: Lungrecruitment manoeuver in prone position.
- Supine position (Active Comparator): Intervention: Lungrecruitment in supine position. Device: Ventilator Flow-i, Peak inspiratory pressure 40 cmH2O, PEEP 20 cm H2O during 30 s. Clinical routine.
  Interventions: Procedure: Lungrecruitment manoeuver in supine position.

INTERVENTIONS:
Procedure: Lungrecruitment manoeuver in prone position. — Postoperative lungrecruitment in prone position, pressure-controlled ventilation peak inspiratory pressure 40 cm H2O combined with PEEP 20 cm H2O during 60 seconds.
  Other Names: "Prone Lungrecruitment in ventilator"
  Arms: Prone position
Procedure: Lungrecruitment manoeuver in supine position. — Postoperative lungrecruitment in supine position, pressure-controlled ventilation peak inspiratory pressure 40 cm H2O combined with PEEP 20 cm H2O during 60 seconds.
  Other Names: "Supine Lungrecruitment in ventilator"
  Arms: Supine position

SUMMARY:
The study comprises two different objectives. Longitudinal description of postoperative pulmonary dysfunction in the cardiothoracic surgery patient, and the comparison of two different lungrecruitment strategies.

DETAILED DESCRIPTION:
Introduction:

Atelectasis and consolidation of lung tissue is a well recognized clinical scenario following anaesthesia, musclerelaxation and mechanical ventilation. In cardiac surgery during cardiopulmonary bypass (CPB), the lungs are collapsed to a degree depending on surgical opening of the pleura, time on bypass, and gasmixture on termination of ventilation. Recruitment of the lungs on commencement of mechanical ventilation after CPB generally must be repeated before extubation. There are several different approaches to Recruitment Manoeuvers (RM). Increasing pressures in the ventilator (peak-pressures and PEEP), increasing tidal volumes and inspiratory hold are facilities offered by the ventilator. Different body positions by interaction of the abdomen and thorax through the diaphragm, and the action of gravity on the lungs and adjoining organs, are other principles. The contribution of spontaneous ventilatory efforts also play a major roll.

Study rationale:

The study comprises two different objectives. Longitudinal description of postoperative pulmonary dysfunction in the cardiothoracic surgery patient, and the comparison of two different lungrecruitment strategies.

All patients undergoing cardiothoracic surgery develops some degree of postoperative pulmonary dysfunction (PPD), including hypoxemia, increased work of breathing, shallow respiration and ineffective cough. Respiratory symptoms of larger clinical significance are better investigated, known as postoperative pulmonary complications (PPC), including pleural effusion, atelectasis, pneumonia and ARDS. Pathophysiology is complex and multifactorial, and there is a continuum between PPD and PPC that has not yet been well explored. A large proportion of patients readmitted to CICU present respiratory failure, significantly accounting for morbidity, mortality, and costs.

Regarding lungrecruitment, supine position is compared to modified prone position with similar ventilator settings. Initial measurements preoperatively in the awake patient, then during sedation and ventilator treatment, followed up by measurements before discharge from the surgical ward on postoperative day 4-5.

Effect of RM is evaluated from ventilator measurement of compliance (C), arterial oxygenation and P/F-ratio from the arterial blood gas (ABG), and electrical impedance tomography (EIT). EIT measures the impedance of a thoracic sagittal section by emitting and sampling electrical currents between 16 electrodes fixed on a submamillar belt. Radiology report from routine chest X-ray and ultrasonography of the lungs and pleura will be added.

Should RM in prone position prove to be more efficient, postoperative complications in terms of respiratory failure and pneumonia could be reduced, facilitating postoperative recovery and shortening convalescens. This would justify the increased burden of care in the cardiac ICU.

Study objectives:

The study aims to compare lung recruitment in two different body positions, supine (elevated 30 degrees) to left modified prone position (left side up, 120 degrees). Parameters investigated are global and regional pulmonary impedance (EIT), lungcompliance, and arterial oxygenation. Chest X-ray and lung ultrasound will be performed for additional analyses.

A descriptive longitudinal study of the 20 patients lungrecruited in supine position will also be performed.

Study design:

Prospective, randomized clinical trial. Two groups with 20 cardiac surgery patients in each.

Study procedure:

Protocol

Day -1:

1 day preop. EIT measurement in supine (30 degrees elevated) and modified left prone position (left side up, 120 degrees). Two measurements of each 2 min duration in both positions. ABG is performed after breathing through a Venturi-mask delivering FiO2 0.5 for 10 minutes. Randomization to either of the two groups.

Day 0:

Day of surgery. Standard periop care in coherence with department routines. Preoxygenation using FiO2 1.0 during induction of anaesthesia, and before commencing cardiopulmonary bypass (CPB). Inhalational anaesthetics during surgical preparation, and again after weaning from CPB. Apnoea without PEEP or intermittent ventilation during CPB. Before weaning from CPB manual lung recruitment with the APL-valve set to 30 cm H2O, and visual guidance of the lungparenchyma or pleura. After chest closure, FiO2 is set to 0.5, volume controlled ventilation 4-6 ml/Kg titrated according to pCO2, and PEEP is set to 5 cm H2O. Patient ventilation circuit will be broken twice in conjugation with the use of a transport ventilator device before arrival in the CICU. Ventilator settings in the CICU is pressure-regulated volume-controlled ventilation (VKTS), tidal volumes of 4-6 ml/Kg titrated according to pCO2, respiratory frequency of 14/min, and PEEP 8 cm H2O.

Recruitment maneuver (RM) is performed within 10 min on arrival in the CICU. Patient must be stabile in hemodynamic parameters, including volume status. PEEP is set to 20 cm H2O, pressure controlled ventilation with peak pressure 40 cm H2O for 30 s (5 inspirations), thereafter PEEP-trial starting from 15 cm H2O for optimal PEEP using the "Open Lung Tool" (Maquet Flow-i software). During the PEEP-trial, VKTS for tidal volumes of 6 ml/Kg is used.

Supine position group: RM in supine position. EIT, ABG and lung compliance measurements in supine position before RM (30 degrees elevation), then immediately and 30 min after RM, and again 30 minutes after extubation. FiO2 0.5 at all ABG measuring points.

Modified prone position group: RM in modified prone position (120 degrees, left side up). EIT, ABG and lung compliance measurements in supine position before RM (30 degrees elevation), and then immediately after RM when turned back to supine position (30 degrees elevation), and 30 minutes after RM. Finally, measurements 30 minutes after extubation. FiO2 0.5 at all ABG measuring points.

Day 4-5:

Supine and prone position groups: EIT in supine position (30 degrees elevation) and ABG repeated at day 4-5 postop. ABG is performed after breathing through a Venturi-mask delivering FiO2 0.5 for 10 minutes. Ultrasonography of the pleurae. Chest-X-ray performed routinely on the day after chest-drain removal.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Scheduled cardiac surgery (CABG or valve surgery)
* Cardiopulmonary bypass

Exclusion Criteria:

* Diagnose of obstructive or restrictive lung disease
* Medical therapy with bronchodilators
* Smoking or former smoking > 5 years
* Obesity (BMI > 30)
* Perioperative FiO2 >60% or PEEP >12
* Haemodynmic instability, use of inotropes (low dose vasopressors accepted)
* Postop clinically significant bleeding (>100 ml/h, reoperation)
* Postoperative haemothorax or large pleural effusion detected with ultrasonography
* Postoperative clinically significant pneumothorax or large chestdrain airleak

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Electrical impedance | 5 days
  Electrical impedance tomography, thoracical transverse plane measurment. Dräger Pulmovista device is used for collecting the data. Data will be transferred to a personal computer, and processed in Excel.
Lungcompliance (ml/cm H2O) | 2 hours
  Pulmonary dynamic compliance, ventilator measurment.
P/F ratio | 5 days
  Oxygenation ratio, pO2 divided by FiO2, indication of pulmonary shunt
Ultrasonography | 5 days
  Lungultrasound to exclude pleural effusion.
Chest X-ray | 5 days
  Chest X-ray to exclude pneumothorax

OTHER OUTCOMES:
Safety and Tolerability of prone position (turned 180 dgrees from supine position, Intensive Care Unit Bed), number of adverse events observed by the primary investigator. | 2 hours
  Placing a patient in prone position in the immediate postoperative and sedated setting in the Cardiac Intensive Care Unit. Adverse events will be observed and noted by the primary investigator. Adverse events will be divided in less severe (e.g disruption of monitoring, uncoupling of breathing curcuit) and severe (e.g accidental extubation, decubitus ulcers, emergency return to supine position).

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Study Chair — The Salgrenska Academy
Locations (1):
- Department of cardiothoracic anaesthesia, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinsson A, Houltz E, Wallinder A, Magnusson J, Lindgren S, Stenqvist O, Thoren A. Inspiratory and end-expiratory effects of lung recruitment in the prone position on dorsal lung aeration - new physiological insights in a secondary analysis of a randomised controlled study in post-cardiac surgery patients. BJA Open. 2022 Nov 21;4:100105. doi: 10.1016/j.bjao.2022.100105. eCollection 2022 Dec. PMID 37588783
- [Derived] Martinsson A, Houltz E, Wallinder A, Lindgren S, Thoren A. Lung recruitment in the prone position after cardiac surgery: a randomised controlled study. Br J Anaesth. 2021 May;126(5):1067-1074. doi: 10.1016/j.bja.2020.12.039. Epub 2021 Feb 16. PMID 33602580